CLINICAL TRIAL: NCT04944966
Title: Evaluation of Safety and Efficacy of Maytenus Senegalensis for the Treatment of Uncomplicated Malaria Episodes in Adult Patients as Compared to Artemether-lumefantrine
Brief Title: Safety and Efficacy of Maytenus Senegalensis for the Treatment of Uncomplicated Malaria
Acronym: MALHERBAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ifakara Health Institute (Other)
Collaborators: Swiss Tropical & Public Health Institute (Other); Muhimbili University of Health and Allied Sciences (Other); National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MALHERBAL
Record Dates: First submitted 2021-05-16; First posted 2021-06-30 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): • Experimental: Group 1a: n=3, Healthy male participants will receive Maytenus senegalensis administered orally at an estimated dose of 400mg once a day to test its safety and tolerability.
  Interventions:
  o Drugs: Maytenus senegalensis
  • Experimental: Group 1b: n=3, Healthy male participants will receive Maytenus senegalensis administered orally at an estimated dose of 600mg once a day to test its safety and tolerability.
  Interventions:
  o Drugs: Maytenus senegalensis
  • Experimental: Group 1c: n=3, Healthy male participants will receive Maytenus senegalensis administered orally at an estimated dose of 800mg for 8 hourly for 4 days to test its safety and tolerability.
  Interventions:
  o Drugs: Maytenus senegalensis
  • Experimental: Group 1d: n=3, Healthy male participants will receive Maytenus senegalensis administered orally at an estimated dose of 800mg for 8 hourly for 4 days to test its safety and tolerability.
  Interventions:
  o Drugs: Maytenus senegalensis
  Interventions: Drug: Maytenus Senegalensis
- Group 2a (Experimental): Group 2a: n=52, Adults aged 18 to 45 years diagnosed with natural acquired uncomplicated malaria will be treated with Maytenus senegalensis.
  Patients will be treated with Maytenus senegalensis administered orally at an estimated dose of 800mg for 8 hourly for 4 days.
  Curative efficacy will be assessed by measure the portion of patients with Early Treatment Failure (ETF), Asexual parasite clearance time (PCT) and adequate Clinical and Parasitological Response (ACPR) for treatment at 28 days and 56 days after PCR correction of reinfection (ACPR 28 and 56 after PCR correction of reinfection
  Interventions:
  o Drugs: Maytenus senegalensis
  Interventions: Drug: Maytenus Senegalensis
- Group 2b (Active Comparator): Group 2a: n=52, Adults aged 18 to 45 years diagnosed with natural acquired uncomplicated malaria will be treated with Artemether-lumefantrine Patients will be treated with Artemether 20mg/lumefantrine 120mg administered orally by a six-dose regimen over 3 days.
  Curative efficacy will be assessed by measure the portion of patients with Early Treatment Failure (ETF), Asexual parasite clearance time (PCT) and adequate Clinical and Parasitological Response (ACPR) for treatment at 28 days and 56 days after PCR correction of reinfection (ACPR 28 and 56 after PCR correction of reinfection
  Interventions:
  o Drugs: Artemether 20mg/lumefantrine 120mg
  Interventions: Drug: Maytenus Senegalensis

INTERVENTIONS:
Drug: Maytenus Senegalensis — * Maytenus senegalensis (Malherbal) has a very long history of safe medicinal use in Africa in adult as well as infants and children. It will be administered orally at a dose of 800mg 8 hourly for 4 days.
  * Artemether 20mg/lumefantrine 120mg
  Other Names: Artemether-lumefantrine

SUMMARY:
Antimalarial Herbal medicine known as Maytenus senegalensis will be evaluated for its safety, tolerability and efficacy among Tanzanian male adults aged 18 to 45 years. The first primary objective is to assess the safety and tolerability of malaria herbal remedy of Maytenus senegalensis among healthy male adults aged 18 to 45 years in Tanzania. And the second objective is to evaluate the safety, tolerability as well as efficacy of malaria herbal remedy Maytenus senegalensis (MALHERBAL) for the treatment of Tanzanian adults aged 18 to 45 years with uncomplicated malaria compared to Artemether-lumefantrine.

DETAILED DESCRIPTION:
The herbal medicine (Maytenus senegalensis) has been scientifically investigated for acute toxicity in vitro and antiplasmodial activity both in vitro and in vivo where it showed strong antimalarial activity. However, to our knowledge, no antimalarial studies have been performed on this herbal medicine in standardized clinical settings.

The study will contain two treatment groups. Group 1 will have 12 healthy male adults aged 18 to 45 years who will be given the malaria herbal remedy (Maytenus senegalensis) and followed up for safety for 56 days. The subgroup 1a will be the first group to be enrolled in the study and given Malaria herbal remedy. The safety assessment of this group will be done in 7 days after the first treatment. If there will be no major safety concern per-protocol among participants of group 1a, the subgroup 1b participants will be enrolled in the study and given Malaria herbal remedy. The safety assessment of this subgroup 1b will be done 7 days after the first treatment. If there will be no major safety concern per-protocol among participants of group 1b, the subgroup 1c participants will be enrolled in the study and given Malaria herbal remedy. The safety assessment of this subgroup 1c will be done 7 days after the first treatment. If there will be no major safety concern per-protocol among participants of group 1c, the subgroup 1d participants will be enrolled in the study and given Malaria herbal remedy. The decision to proceed from G1 to the enrolment of G 2 participants will be determined by pre-specified "go or no go" criteria.

Study group 2 will comprise two subgroups of male Adults aged 18 to 45 years with uncomplicated malaria. The first is study group 2a of 52 uncomplicated malaria patients who will be treated with the malaria herbal remedy (Maytenus senegalensis) while G2b of 52 uncomplicated malaria patients will be treated with Artemether-lumefantrine. Patients will be followed up for 56 days. In the presence of failure for either the herbal remedy and Artemether-lumefantrine and Early Treatment Failure criteria met, the rescue treatment will be used.

The purpose of utilizing Group 1 participants is to assess the safety and tolerability of Maytenus senegalensis and proof of the concept that the herbal product is safe for the human subject. Therefore, the decision to proceed to Group 2 intervention for patients with naturally acquired malaria will be subjected to pre-specified "go or no go" criteria. These criteria will be based on safety data obtained from the sentinel group of 12 participants on day 28 after the first treatment and will be reviewed by an independent safety monitoring committee (SMC) appointed for this study. If one of the following criteria will be met, the study will not enroll the remaining G2 participants: (i)Any SAE related to the antimalarial herbal remedy (ii) ≥50% of the participants experienced a Grade 3 AR persisting at Grade 3 for > 48 hours during the 14 follow-up days.

ELIGIBILITY:
Group 1

Inclusion Criteria:

* Healthy males based on clinical and laboratory findings
* Aged from 18 to 45 years
* Adults with a Body Mass Index (BMI) 18 to 30 Kg/m2.
* Long-term (at least one year) or permanent residence in the Bagamoyo district or nearby districts.
* Agreement to release medical information and to inform the study doctor concerning contraindications for participation in the study.
* Willingness to be attended to by a study clinician and take all necessary medications prescribed during the study period
* Agreement to provide contact information of a third-party household member or close friend to study team
* Availability through mobile phone 24 hours during the entire study period
* Agreement not to participate in another clinical trial during the study period
* Agreement not to donate blood during the study period
* Able and willing to complete the study visit schedule over the study follow up period, including the hospitalizations required for protocol compliance
* Willingness to undergo HIV, hepatitis B (HBV) and hepatitis C (HCV) tests
* Able to demonstrate their understanding of the study by responding correctly to 10 out of 10 true/false statements (in a maximum of two attempts for those who failed to respond correctly to all true/false statements in the first attempt)
* Signed written informed consent, in accordance with local practice
* Free from malaria parasitaemia by blood smear at enrolment

Exclusion Criteria:

* Previous receipt of an investigational malaria drug in the last 5 years
* Participation in any other clinical study involving investigational medicinal products within 30 days prior to the onset of the study or during the study period
* History of arrhythmias or prolonged QT-interval or another cardiac disease, or clinically significant abnormalities in electrocardiogram (ECG) at screening
* Positive family history in a 1st or 2nd-degree relative for the cardiac disease at age <50 years old
* A history of psychiatric disease
* Suffering from any chronic illness including; diabetes mellitus, cancer or HIV/AIDS
* Any confirmed or suspected immunosuppressive or immune-deficient condition, including asplenia
* History of drug or alcohol abuse interfering with normal social function
* The use of chronic immunosuppressive drugs or other immune-modifying drugs within three months of study onset except inhaled and topical corticosteroids.
* Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis
* Positive HIV, hepatitis B virus or hepatitis C virus tests
* Suspected of having clinically active TB by history or physical examination with positive QuantiFERON-TB Gold Test In-Tube assay
* Symptoms, physical signs and laboratory values suggestive of systemic disorders including renal, hepatic, blood, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, and other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteers.
* Any medical, social condition, or occupational reason that, in the judgment of the study clinician, is a contraindication to protocol participation or impairs the volunteer's ability to give informed consent, increases the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data

Group 2

Inclusion Criteria:

* Male adults aged from 18 to 45 years
* Ability to swallow oral medication
* Adults with a Body Mass Index (BMI) 18 to 30 Kg/m2.
* Uncomplicated malaria, with microscopically confirmed mono-infection by P. falciparum (parasitaemia ≥1.000/ μL and <200,000/ μL).
* History of fever anytime during the preceding 24 hours or presence of fever (axillary temperature ≥37.5 °C or rectal ≥38.0 °C).
* Ability to understand the nature of the trial
* Ability and willingness to comply with the protocol for the duration of the study, study visit schedule and to provide informed consent from.
* Stable residence in the study area during the two months after recruitment.

Exclusion Criteria:

* A history of antimalarial drug use such as Amodiaquine, Chloroquine, Quinine or lumefantrine-based compounds within the previous 6 weeks, with Piperaquine-based compound, or Mefloquine, or Sulphadoxine/pyrimethamine (SP) within the previous 3 months and with Halofantrine within the 30 days prior to screening.
* Any other antimalarial drug or antibiotics use with antimalarial activity (including cotrimoxazole) and any herbal products, within the 7 days prior to screening.
* Presence of any febrile condition due to severe diseases other than malaria (e.g. measles, pneumonia, typhoid fever, UTI, meningitis
* Presence of general danger signs or signs of severe falciparum malaria according to the definitions of WHO
* Known hypersensitivity to the artemisinin-based therapy.
* History of the relevant clinical allergic reaction of any origin.
* Known moderate/ severe renal or liver insufficiency.
* Evidence of clinically relevant hematological, pulmonary, metabolic-endocrine, neurological, urogenital diseases as judged by the study clinician.
* Suffering from any chronic illness including; cancer or HIV/AIDS or hepatitis B virus (HBV) or HCV infection
* Previous admission for, or evidence of symptomatic cardiac arrhythmias or with clinically relevant bradycardia at screening (bpm < 40).
* Family history of sudden death, or known congenital prolongation of the QT interval, or any clinical condition known to prolong the QT interval.
* Any other ECG abnormality that requires urgent management.
* Gastrointestinal dysfunction that could alter absorption or motility (i.e. malabsorption syndromes, intestinal sub occlusion or previous major gastrointestinal surgery).
* Any clinically significant deviation from the normal range in biochemistry or hematology blood tests or in urine analysis
* Severe anemia (Hb < 7.9 g/dL).
* Participation in any investigational drug study during the 42 days prior to screening

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2022-09-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinical significance abnormal values in hematology parameters during the follow up period of 28 days for all participants of group 1 and 2. | up period of 28 days
  Blood samples will be collected for the analysis of hematology parameters including Red cell blood count (RBC), hemoglobin (HBG), platelets (PLT), white blood cell count (WBC) with differential (neutrophil (NEUT), lymphocyte (LYMPH), and eosinophil (EO)) counts. Blood sample will be collected at Day 0(Baseline), Day 3, day 7, Day 14 and Day 28 Clinical significance abnormal values hematology parameter will be determined by adapted FDA Toxicity Grading Scale.
Number of participants with clinical significance abnormal values in biochemistry parameters during the follow up period of 28 days for all participants of group 1 and 2. | up period of 28
  Blood samples will be collected for the analysis of biochemistry parameters including ASAT, bilirubin total and creatinine. Blood sample will be collected at Day 0(Baseline), Day 3, day 7, Day 14 and Day 28. Clinical significance abnormal values of Biochemistry parameters will be determined by adapted FDA Toxicity Grading Scale.
Number of participants with significant changes in vital signs comparing to baseline during the follow up period of 28 days for all participants of group 1 and 2. | up period of 28
  Vital signs assessment included heart rate (HR), systolic blood pressure (SBP) and diastolic blood pressure (DBP). Assessments were completed at Day 0 (Baseline), Day 1 up to Day 7, Day 14, and Day 28. We be reviewed using locally prepared normal range for vital sign
Number of AEs during the follow up period of 28 days for all participants of group 1 and 2 | up period of 28
  An Adverse Event is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The analysis was performed on all participants who received at least one dose of study treatment.
Number of SAEs during the follow up period of 56 days for all participants of group 1 and 2 | Up period of 56
  SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/ incapacity, other situations and is associated with liver injury or impaired liver function. The analysis was performed on all participants who received at least one dose of study treatment.
Number of participants of group 2 with Early Treatment Failure (ETF), | Day 1 up to 3
  Development of danger signs or severe malaria on Day 1, Day 2 or Day 3 in the presence of parasitaemia, parasitaemia on Day 2 higher than on Day 0, irrespective of axillary temperature, parasitaemia on Day 3 with axillary temperature ≥ 37.5 ºC and parasitaemia on Day 3 ≥ 25% of count on day 0.
Number of participants of group 2 with Late Treatment Failure (LTF) | Day 4 up to 28
  Development of danger signs or severe malaria on any day from day 4 to day 28 in the presence of parasitaemia; without previously meeting any of the criteria of Early Treatment Failure; Presence of parasitemia + axillary temperature ≥37.5°C on any day from Day 4 to Day 28, without previously meeting any criteria of ETF.
Number of participants of group 2 with Late parasitology failure (LPF) | Day 7-28
  Presence of parasitemia on any day from D7 to D28 + axillary temperature <37.5°C, without previously meeting any of the criteria of ETF

SECONDARY OUTCOMES:
Number of participants of group 2 with Adequate Clinical and Parasitological Response (ACPR) | 28 days
  Absence of parasitaemia on day 28 irrespective of axillary temperature without previously meeting any of the criteria of Early Treatment Failure or Late Clinical Failure or Late Parasitological Failure.

OTHER OUTCOMES:
Number of developed early ring stage P. falciparum parasites | Day 0,3,14 and 28
  A blood sample for in vitro drug testing will be collected from the participants of study group 2b on days 0, 3, 14 and 28 in order to evaluate in vitro susceptibility of P. falciparum isolates to Artemether-lumefantrine (Determination of early ring stage of P. falciparum)
Percentage of inhibitory concentration (IC50 and IC90) values of the Artemether-lumefantrine | Day 0,3,14 and 28
  A blood sample for in vitro drug testing will be collected from the participants of study group 2b on days 0, 3, 14 and 28 in order to evaluate in vitro susceptibility of P. falciparum isolates to Artemether-lumefantrine
Percentage of identified resistance molecular marker of Artemether-lumefantrine | Day 0,3,7,14,28 and 56
  Two to three drops of blood will be collected on filter paper from the participants of study Group 2b on days 0, 3, 7, 14, 28 and 56 to study the polymorphism or copy number of pfcrt, pfmdr1, pfdhfr and pfdhps genes, which are considered as markers of resistance to Artemether-lumefantrine

CONTACTS AND LOCATIONS:
Overall Officials: Kamaka Kassim, BscN,MPH, Principal Investigator — Ifakara Health Institute
Locations (1):
- Bagamoyo Clinical Trial Facility, Bagamoyo, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kassimu KR, Ali AM, Omolo JJ, Mdemu A, Machumi F, Ngasala B. The effect of an anti-malarial herbal remedy, Maytenus senegalensis, on electrocardiograms of healthy Tanzanian volunteers. Malar J. 2024 Apr 12;23(1):103. doi: 10.1186/s12936-024-04935-w. PMID 38609987